CLINICAL TRIAL: NCT03456388
Title: A Phase ⅠAscending Single-dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Ammoxetine Hydrochloride Enteric-coated Tablets in Chinese Healthy Subjects
Brief Title: Study of Ammoxetine Hydrochloride Enteric-coated Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMXT201701/PRO
Record Dates: First submitted 2017-08-09; First posted 2018-03-07 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ammoxetine Hydrochloride Enteric-coated Tablets (Experimental): There will be 7 ascending cohorts . Each cohort will be administered in different dose once for 7 days.
  Interventions: Drug: Ammoxetine Hydrochloride Enteric-coated Tablets
- Placebo Enteric-coated Tablets (Active Comparator): There will be 7 ascending cohorts. placebo enteric-coate tablets to mimic Ammoxetine Hydrochloride Enteric-coated tablets.
  Interventions: Drug: placebo enteric-coated tablets

INTERVENTIONS:
Drug: Ammoxetine Hydrochloride Enteric-coated Tablets — There will be 7 ascending cohorts. The first cohort will be administered 2.5 mg once. The second cohort will be administered 7.5 mg. The third cohort will be administered 15 mg once. The forth cohort will be administered 30 mg once. The fifth cohort will be administered 45 mg once. The sixth cohort will be administered 65 mg once.The seventh cohort will be administered 100 mg once. The results of each dose group were shown to be safe and tolerable, and then the next dose group was tested.
  Arms: Ammoxetine Hydrochloride Enteric-coated Tablets
Drug: placebo enteric-coated tablets — There will be 7 ascending cohorts. The first cohort will be administered 2.5 mg once. The second cohort will be administered 7.5 mg. The third cohort will be administered 15 mg once. The forth cohort will be administered 30 mg once. The fifth cohort will be administered 45 mg once. The sixth cohort will be administered 65 mg once.The seventh cohort will be administered 100 mg once. The results of each dose group were shown to be safe and tolerable, and then the next dose group was tested.
  Arms: Placebo Enteric-coated Tablets

SUMMARY:
This study evaluates the safety, tolerability and pharmacokinetics of Ammoxetine Hydrochloride Enteric-coated Tablets in Chinese heathy subjects. Part of the participants will receive Ammoxetine Hydrochloride Enteric-coated Tablets, while the other part will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-45 years
* Body weight ≥ 45kg (female) or 50Kg (male), 18 ≤ BMI ≤ 26
* Vital signs, physical examinations and laboratory tests and other tests prove participants are healthy
* Sign the informed consent form voluntarily and cooperate voluntarily to complete the test

Exclusion Criteria:

* Allergens (allergic to 2 or more drugs, food or pollen)
* comorbid illness (mental illness, liver and kidney disease, gastrointestinal diseases, nervous system disease, or other systemic diseases)
* have Clinically significant abnormal screening laboratory values.
* Systolic pressure > 140mmHg or diastolic > 90 mmHg
* Postural hypotension (systolic blood pressure drop by 20mmHg or diastolic blood pressure drop by 10mmHg after standing position)
* The QTc period ≥ 450ms (male) or 470ms (female) or has a history of QTc extension
* Smoking or alcohol consumption (14 units per week in the previous 4 weeks : 1 unit = beer 285mL, or 25mL of spirits, or 150 mL of wine; Daily smoking ≥ 5) or abusing in past year of drug and other substance
* Have donated blood > 400 ml within 8 weeks prior to screening
* Participated in other clinical trials within 3 months prior to screening
* Intaked too much caffeinated beverage or food within 4 weeks prior to screening. such as: Coffee, tea, chocolate, cola, red bull (no more than 6 units per day). 1 unit of caffeine = 1 cup of coffee (177.4 mL) = 2 pots of cola (354.9 mL) = 1 cup of tea (354.9 mL) = 1/2 cup energy drink = 85g chocolate
* Have taken drugs that changed liver enzyme activity, such as dexamethasone, ketoconazole, rifampicin and omeprazole, were used within 4 weeks prior to screening
* Have taken prescription drugs and OTC (except for the occasional use of acetaminophen and nasal sprays), herbs vitamins or minerals within 4 weeks prior to screening. The interval from prior treatment to screening should be at least 5 half-lives metablism which subjected to the longer half-life
* Using any psychotropic drug or psychoactive substance
* Women were screened for positive blood pregnancy
* The subjects and their partners were not willing to take contraceptives during trial and six months after the study
* Have a donor plan recently
* Have participated in this trial
* The researchers believe that anyone who is unfit to participate in this test will be involved

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 8 days
  Incidence of Adverse Events that researchers determined clinical significance

SECONDARY OUTCOMES:
Pharmacokinetics of blood sample | 8 days
  changes in blood concentration
Mass balance | 8 days
  the metabolite analysis in sample of plasma, urine and fecal.
Pharmacokinetics of urine sample | 8days
  changes in urine concentration

CONTACTS AND LOCATIONS:
Overall Officials: Qi Shen, Principal Investigator — Sichuan huaxi hospital 1 ward.
Locations (1):
- Sichuan huaxi hospital 1 ward., Chengdu, Sichuan, China